CLINICAL TRIAL: NCT01987817
Title: Phase 2 Oral Desensitization to Peanut in Peanut-Allergic Children and Adults Using Characterized Peanut Allergen Oral Immunotherapy
Brief Title: Oral Desensitization to Peanut in Peanut-Allergic Children and Adults Using Characterized Peanut Allergen OIT
Acronym: ARC001
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aimmune Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ARC001
Record Dates: First submitted 2013-11-13; First posted 2013-11-19 (Estimated); Results first posted 2021-11-02 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Peanut Allergy
Keywords: Characterized Peanut Allergen; Peanut; OIT; Oral Desensitization; Peanut Allergen; Allergy; Peanut Allergy; Peanut-Allergic Children; Children; Peanut-Allergic Adults
MeSH Terms: conditions — Peanut Hypersensitivity; Hypersensitivity | interventions — Capsules

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AR101 powder provided in capsules (Experimental): Study product provided as peanut protein in pull-apart capsules
  Interventions: Biological: AR101 powder provided in capsules
- Placebo powder provided in capsules (Placebo Comparator): Placebo formulation in pull-apart capsules containing only inactive ingredients
  Interventions: Biological: Placebo powder provided in capsules

INTERVENTIONS:
Biological: AR101 powder provided in capsules — Study product formulated to contain peanut protein at different dosage strengths for use as defined in the protocol
  Arms: AR101 powder provided in capsules
Biological: Placebo powder provided in capsules — Study product formulated to contain only inactive ingredients for use as defined in the protocol
  Arms: Placebo powder provided in capsules

SUMMARY:
This is a multi-center, randomized, double-blind placebo controlled study of efficacy and safety of characterized peanut oral immunotherapy in peanut allergic individuals.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind placebo controlled study of efficacy and safety of characterized peanut OIT in peanut allergic individuals. All eligible subjects will receive an escalating dose of CPNA or placebo. Approximately 50 subjects will be randomized 1:1 to peanut OIT or placebo.

ELIGIBILITY:
Key Inclusion Criteria:

* Ages 4 through 26 years, inclusive
* Clinical history of allergy to peanuts or peanut-containing foods
* Serum IgE to peanut >0.35 kU/L (determined by UniCAP within the past 12 months) and/or a SPT to peanut >3 mm compared to control
* Experience dose-limiting symptoms at or before the 100mg dose of peanut protein (measured as 200 mg of peanut flour) on abbreviated screening OFC conducted via PRACTALL guidelines
* Use of birth control by females of child-bearing potential

Key Exclusion Criteria:

* History of Cardiovascular disease
* History of frequent or repeated, severe or life-threatening episodes of anaphylactic shock
* History of other chronic disease
* History of eosinophilic gastrointestinal disease
* Severe asthma
* Mild or moderate asthma if uncontrolled
* Use of omalizumab within the past 6 months or current use of other non-traditional forms of allergen immunotherapy
* Use of beta-blockers(oral), angiotensin-converting enzyme (ACE)
* Pregnancy, lactation
* Having the same place of residence as another study subject
* Participation in an interventional clinical trial 30 days prior to randomization

Ages: 4 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 56 (Actual)
Dates: Start 2014-02-06 (Actual); Primary Completion 2015-01-07 (Actual); Study Completion 2015-01-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Director of Regulatory Affairs, Study Chair — Aimmune Therapeutics, Inc.
Locations (8):
- United States (8):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - UC San Diego, San Diego, California
  - Boston Children's Hospital, Boston, Massachusetts
  - Mount Sinai Medical Center, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Medical Center Dallas, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nilsson C, Scurlock AM, Dellon ES, Brostoff JM, Pham T, Ryan R, Brown KR, Adelman DC, Aceves SS. Onset of eosinophilic esophagitis during a clinical trial program of oral immunotherapy for peanut allergy. J Allergy Clin Immunol Pract. 2021 Dec;9(12):4496-4501. doi: 10.1016/j.jaip.2021.07.048. Epub 2021 Aug 11. No abstract available. PMID 34389504

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 67 subjects signed the informed consent and went through the screening process. 11 subjects failed screening, resulting in 56 subjects being enrolled and initially randomized. The randomized population comprised 29 subjects in the AR101 group and 27 subjects in the placebo group. The final intent-to-treat (ITT) population (subjects who received at least 1 dose of randomized study treatment) had one fewer subject in the placebo group (n=26).
Period: Overall Study
Arm/Group | AR101 Powder Provided in Capsules | Placebo Powder Provided in Capsules
Started | 29 | 27
Completed | 23 | 26
Not Completed | 6 | 1
Not completed — Adverse Event | 4 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: These values reflect the intent-to-treat population (subjects who received at least 1 dose of randomized study treatment)
Groups:
- Total: Total of all reporting groups
Arm/Group | AR101 Powder Provided in Capsules | Placebo Powder Provided in Capsules | Total
Number analyzed (Participants) | 29 | 26 | 55
Age, Continuous [Median (Full Range); unit: years] | 7.0 [4 to 21] | 8.0 [4 to 14] | 8.0 [4 to 21]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 20 | 16 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 29 | 26 | 55
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 26 | 20 | 46
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Subjects Who Tolerate at Least 300 mg (443 mg Cumulative) of Peanut Protein With no More Than Mild Symptoms at the Exit DBPCFC
Description: The primary endpoint was the percentage of subjects who achieved desensitization, as determined by tolerating at least 300 mg (443 mg cumulative) of peanut protein at the Exit Double Blind Placebo Controlled Food Challenge (DBPCFC) with no more than mild symptoms (i.e., desensitization responders)
Time Frame: 6-9 Months
Population: The number of participants analyzed per outcome measure reflects the intent-to-treat (ITT) population (subjects who received at least 1 dose of randomized study treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | AR101 Powder Provided in Capsules | Placebo Powder Provided in Capsules
Number analyzed (Participants) | 29 | 26
Participants | 23 | 5
Statistical Analysis 1: Comparison: AR101 Powder Provided in Capsules vs Placebo Powder Provided in Capsules; Test type: Superiority; p < 0.0001, Fisher Exact; Risk Difference (RD) = 60.0, 95% CI 2-sided [35 to 79]

2. Secondary Outcome: Change From Baseline in Maximum Tolerated Dose of Peanut Protein at the Exit DBPCFC
Description: The change in maximum tolerated dose of peanut protein from baseline (screening) to the Exit Double-Blind, Placebo-Controlled Food Challenge
Time Frame: 6-9 months
Population: The number of participants analyzed per outcome measure reflects the intent-to-treat (ITT) population (subjects who received at least 1 dose of randomized study treatment
Measure: Least Squares Mean (95% Confidence Interval); unit: Change from baseline in MTD (log10 mg)
Arm/Group | AR101 Powder Provided in Capsules | Placebo Powder Provided in Capsules
Number analyzed (Participants) | 29 | 26
Change from baseline in MTD (log10 mg) | 1.254 [0.984 to 1.523] | 0.341 [0.057 to 0.626]
Statistical Analysis 1: Comparison: AR101 Powder Provided in Capsules vs Placebo Powder Provided in Capsules; MTD for the baseline and Exit DBPCFC are transformed back to log10 scale before calculations. A value of 0.3 mg is substituted for subjects who could not tolerate the lowest DBPCFC dose before log10 transformation; Test type: Superiority; p < 0.0001, ANCOVA — The p-value is based on the F-test for treatment effect adjusted for MTD from baseline (log10 mg). The p-value and confidence intervals are based on the normality assumption; Least squares means and 95% CIs based on ANCOVA model of change from baseline in MTD at Exit DBPCFC (terms for treatment & MTD at baseline (log10 mg); Treatment difference = 0.912, 95% CI 2-sided [0.5184 to 1.3065]

3. Secondary Outcome: Number of Participants by Maximum Dose Achieved With no or Mild Symptoms at Exit DBPCFC
Time Frame: 6-9 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | AR101 Powder Provided in Capsules | Placebo Powder Provided in Capsules
Number analyzed (Participants) | 29 | 26
Participants
  0.3 mg | 0 | 1
  3 mg | 2 | 2
  10 mg | 3 | 7
  30 mg | 1 | 5
  100 mg | 0 | 6
  300 mg | 5 | 5
  600 mg | 18 | 0

4. Secondary Outcome: Changes in Peanut-Specific IgE From Baseline to Exit DBPCFC
Time Frame: 6-9 months
Population: The number of participants analyzed per outcome measure reflects the intent-to-treat (ITT) population (subjects who received at least 1 dose of randomized study treatment)
  Relative change from baseline is calculated as the ratio of exit visit result to the baseline result, within treatment group.
Measure: Geometric Mean (95% Confidence Interval); unit: kUA/L
Arm/Group | AR101 Powder Provided in Capsules | Placebo Powder Provided in Capsules
Number analyzed (Participants) | 29 | 26
kUA/L
  Peanut-Specific IgE, Baseline | 32.571 [18.626 to 56.957] | 53.839 [34.952 to 82.934]
  Peanut-Specific IgE, Exit: number analyzed (Participants) | 27 | 26
  Peanut-Specific IgE, Exit | 36.889 [21.258 to 64.015] | 57.060 [37.186 to 87.557]
  Relative Change From Baseline of Peanut-Specific IgGE: number analyzed (Participants) | 27 | 26
  Relative Change From Baseline of Peanut-Specific IgGE | 1.231 [1.027 to 1.475] | 1.060 [1.001 to 1.122]

5. Secondary Outcome: Changes in Peanut-Specific IgG4 From Baseline to Exit DBPCFC
Time Frame: 6-9 months
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | AR101 Powder Provided in Capsules | Placebo Powder Provided in Capsules
Number analyzed (Participants) | 29 | 26
μg/mL
  Peanut-Specific IgG4, Baseline | 0.734 [0.487 to 1.107] | 0.510 [0.344 to 0.757]
  Peanut-Specific IgG4, Exit: number analyzed (Participants) | 28 | 26
  Peanut-Specific IgG4, Exit | 3.609 [2.074 to 6.281] | 0.540 [0.377 to 0.775]
  Relative Change From Baseline of Peanut-Specific IgG4 | 5.068 [3.640 to 7.055] | 1.066 [0.905 to 1.255]

6. Secondary Outcome: Change in Skin Prick Test (SPT) Mean Peanut Wheal Diameter Results From Baseline
Time Frame: Baseline, 6-9 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: millimeter
Arm/Group | AR101 Powder Provided in Capsules | Placebo Powder Provided in Capsules
Number analyzed (Participants) | 29 | 26
millimeter
  Peanut Wheal, Baseline (mm) | 14.1 [11.6 to 16.7] | 13.7 [11.4 to 16.0]
  Peanut Wheal, Exit (mm): number analyzed (Participants) | 28 | 26
  Peanut Wheal, Exit (mm) | 7.1 [5.7 to 8.6] | 11.8 [9.3 to 14.4]
  Change in Peanut Wheel from Baseline (mm): number analyzed (Participants) | 28 | 26
  Change in Peanut Wheel from Baseline (mm) | -7.0 [-9.9 to -4.1] | -1.8 [-4.8 to -1.1]

ADVERSE EVENTS:
Time Frame: 6-9 months
Arm/Group | AR101 Powder Provided in Capsules | Placebo Powder Provided in Capsules
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/26
Serious Adverse Events (participants affected / at risk) | 1/29 | 1/26
Other Adverse Events (participants affected / at risk) | 28/29 | 22/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AR101 Powder Provided in Capsules (N=29) | Placebo Powder Provided in Capsules (N=26)
Hypersensitivity (Immune system disorders) | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AR101 Powder Provided in Capsules (N=29) | Placebo Powder Provided in Capsules (N=26)
Hypersensitivity (Immune system disorders) | 26 | 14
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 5
Viral Infection (Infections and infestations) | 3 | 1
Pharyngitis streptococcal (Infections and infestations) | 2 | 1
Croup Infectious (Infections and infestations) | 1 | 0
Ear infection (Infections and infestations) | 0 | 1
Ear lobe infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0
Molluscum contagiosum (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Otitis externa (Infections and infestations) | 1 | 0
Tinea infection (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 3
Nausea (Gastrointestinal disorders) | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2
Dental caries (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Headache (Nervous system disorders) | 3 | 3
Presyncope (Nervous system disorders) | 1 | 1
Somnolence (Nervous system disorders) | 2 | 0
Dizziness (Nervous system disorders) | 0 | 1
Pyrexia (General disorders) | 5 | 4
Malaise (General disorders) | 0 | 2
Arthropod stings (Injury, poisoning and procedural complications) | 1 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 2
Animal bite (Injury, poisoning and procedural complications) | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 1
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 3 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1
Papule (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 2 | 0
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 1
Conjunctivitis allergic (Eye disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1
Tooth extraction (Surgical and medical procedures) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
* Institutions cannot publish until the multi-center sponsor publication is published
* Or, institutions cannot publish until 18 months after study completion
* And Sponsor review of any publications is required prior to any institution publications according to contractual agreements

DOCUMENTS (2):
  • Study Protocol (2014-05-14): https://cdn.clinicaltrials.gov/large-docs/17/NCT01987817/Prot_000.pdf
  • Statistical Analysis Plan (2015-02-06): https://cdn.clinicaltrials.gov/large-docs/17/NCT01987817/SAP_001.pdf